CLINICAL TRIAL: NCT03611881
Title: Assessing the Integration of Tobacco Cessation Treatment Into Lung Cancer Screening
Brief Title: Assessing the Integration of Tobacco Cessation Treatment Into Lung Cancer Screening (LCS)
Acronym: ScreenASSIST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elyse Park, PhD, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2018P000539/PHS
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Smoking, Tobacco
Keywords: lung screening
MeSH Terms: conditions — Tobacco Smoking | interventions — Counseling; Tobacco Use Cessation Devices; Community Resources

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Short, Short, Present (Experimental): 4 weeks of counseling (by phone or videoconferencing) + 2 weeks of nicotine patch + referral to community resource.
  Interventions: Behavioral: Counseling; Drug: Nicotine patch; Behavioral: Community Resource
- Short, Long, Present (Experimental): 4 weeks of counseling (by phone or videoconferencing) + 8 weeks of nicotine patch + referral to community resource.
  Interventions: Behavioral: Counseling; Drug: Nicotine patch; Behavioral: Community Resource
- Long, Short, Present (Experimental): 8 weeks of counseling (by phone or videoconferencing) + 2 weeks of nicotine patch + referral to community resource.
  Interventions: Behavioral: Counseling; Drug: Nicotine patch; Behavioral: Community Resource
- Long, Long, Present (Experimental): 8 weeks of counseling (by phone or videoconferencing) + 8 weeks of nicotine patch + referral to community resource.
  Interventions: Behavioral: Counseling; Drug: Nicotine patch; Behavioral: Community Resource
- Short, Short, Absent (Experimental): 4 weeks of counseling (by phone or videoconferencing) + 2 weeks of nicotine patch + no referral to community resource.
  Interventions: Behavioral: Counseling; Drug: Nicotine patch
- Short, Long, Absent (Experimental): 4 weeks of counseling (by phone or videoconferencing) + 8 weeks of nicotine patch + no referral to community resource.
  Interventions: Behavioral: Counseling; Drug: Nicotine patch
- Long, Short, Absent (Experimental): 8 weeks of counseling (by phone or videoconferencing) + 2 weeks of nicotine patch + no referral to community resource.
  Interventions: Behavioral: Counseling; Drug: Nicotine patch
- Long, Long, Absent (Experimental): 8 weeks of counseling (by phone or videoconferencing) + 8 weeks of nicotine patch + no referral to community resource.
  Interventions: Behavioral: Counseling; Drug: Nicotine patch

INTERVENTIONS:
Behavioral: Counseling — 4 or 8 weeks of behavioral counseling support to promote smoking cessation.
Drug: Nicotine patch — 2 or 8 weeks of nicotine patch given in a tapering dose of 21 mg, 14 mg, 7 mg.
  Other Names: NRT
Behavioral: Community Resource — Counselor-facilitated referral to a community-based program to address social needs.
  Arms: Long, Long, Present; Long, Short, Present; Short, Long, Present; Short, Short, Present

SUMMARY:
This randomized controlled trial seeks to evaluate the effectiveness of alternative strategies to integrate smoking cessation interventions into the delivery of low-dose CT (LDCT) lung cancer screening. Using a factorial design, current smokers who enroll will be randomly assigned to receive these interventions: (1) smoking cessation counseling support by telephone or videoconferencing (short duration vs. long duration); (2) nicotine patch treatment (NRT) (short vs.long duration); (3) counselor-facilitated referral (vs. no referral) to an online resource to connect smokers to a community-based social service resources.

DETAILED DESCRIPTION:
Evidence-based tobacco dependence treatment consists of behavioral counseling and pharmacotherapy. Nicotine patch is an FDA-approved cessation aid. The optimal duration of counseling and pharmacotherapy for patients undergoing low-dose CT (LDCT) lung screening is not clear. In addition, helping smokers to address other social and psychological barriers might help them succeed in quitting smoking. This randomized controlled trial will test, in a factorial design, two options for delivering each of 3 interventions to help current smokers stop smoking in the context of having routine CT lung cancer screening. Patients will receive 4 or 8 weeks of behavioral counseling (with their choice of video conferencing or regular telephone calls), 2 or 8 weeks of nicotine patch, and will receive referral (vs. no referral) to an online resource to connect smokers to community-based social service resources. Outcome measures for smoking cessation will be assessed by a survey administered by phone at 3,and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo LDCT-LCS at a participating Mass General Brigham Health Care System LCS site
* Speak English or Spanish.
* Current smokers: smoked a cigarette, even a puff, in the last 30 days.
* Medicare coverage requirement (age 50-80 years, 20+ pack/years).
* Residing within the USA.

Exclusion Criteria:

* Undergoing lung CT as part of a diagnostic or abnormal follow-up evaluation.
* Unable to give informed consent due to psychiatric or cognitive impairment as determined in consultation with study PI or treating clinician.
* No access to a telephone or cannot communicate by telephone.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elyse R Park, PhD, Principal Investigator — Massachusetts General Hospital; Nancy A Rigotti, MD, Principal Investigator — Massachusetts General Hospital; Jennifer Haas, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Brigham & Women's Faulkner Hospital, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Martha's Vineyard Hospital, Oak Bluffs, Massachusetts
  - Salem Hospital, Salem, Massachusetts

REFERENCES:
- [Derived] Park ER, Haas JS, Rigotti NA, Neil JM, Marotta CJ, Wint AJ, Gonzalez I, McGovern SE, Chang Y, Levy DE, Flores EJ, Merker VL, Noonan E, Bliss CC. Integrating Tobacco Treatment Into Lung Cancer Screening: The Screen Assist Factorial Randomized Clinical Trial. JAMA Intern Med. 2025 May 1;185(5):531-539. doi: 10.1001/jamainternmed.2024.8399. PMID 40029643
- [Derived] Park ER, Neil JM, Noonan E, Howard SE, Gonzalez I, Marotta C, Wint AJ, Levy DE, Chang Y, Rigotti NA, Haas JS. Leveraging the Clinical Timepoints in Lung Cancer Screening to Engage Individuals in Tobacco Treatment. JNCI Cancer Spectr. 2022 Nov 1;6(6):pkac073. doi: 10.1093/jncics/pkac073. PMID 36350049

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Short, Short, Present | Short, Long, Present | Long, Short, Present | Long, Long, Present | Short, Short, Absent | Short, Long, Absent | Long, Short, Absent | Long, Long, Absent
Started | 82 | 82 | 80 | 79 | 79 | 81 | 81 | 78
Completed | 82 | 82 | 80 | 79 | 79 | 81 | 81 | 78
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Short, Short, Present | Short, Long, Present | Long, Short, Present | Long, Long, Present | Short, Short, Absent | Short, Long, Absent | Long, Short, Absent | Long, Long, Absent | Total
Number analyzed (Participants) | 82 | 82 | 80 | 79 | 79 | 81 | 81 | 78 | 642
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 49 | 40 | 47 | 50 | 45 | 49 | 48 | 377
  >=65 years | 33 | 33 | 40 | 32 | 29 | 36 | 32 | 30 | 265
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 43 | 40 | 47 | 48 | 51 | 50 | 35 | 358
  Male | 38 | 39 | 40 | 32 | 31 | 30 | 31 | 43 | 284
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 5 | 6 | 2 | 8 | 7 | 7 | 47
  Not Hispanic or Latino | 75 | 73 | 73 | 72 | 70 | 69 | 72 | 67 | 571
  Unknown or Not Reported | 2 | 2 | 2 | 1 | 7 | 4 | 2 | 4 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 6
  Asian | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 14 | 6 | 10 | 9 | 8 | 7 | 6 | 7 | 67
  White | 65 | 72 | 67 | 63 | 70 | 68 | 70 | 65 | 540
  More than one race | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 5
  Unknown or Not Reported | 2 | 2 | 1 | 4 | 0 | 3 | 4 | 5 | 21
Language [Count of Participants; unit: Participants]
  English | 78 | 80 | 79 | 76 | 78 | 77 | 78 | 75 | 621
  Spanish | 4 | 2 | 1 | 3 | 1 | 4 | 3 | 3 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Self-reported Past 7-day Smoking Abstinence
Description: Number of participants that self-reported no cigarette smoking in the past 7 days
Time Frame: 6 Months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Short, Short, Present | Short, Long, Present | Long, Short, Present | Long, Long, Present | Short, Short, Absent | Short, Long, Absent | Long, Short, Absent | Long, Long, Absent
Number analyzed (Participants) | 82 | 82 | 80 | 79 | 79 | 81 | 81 | 78
Participants | 12 | 10 | 12 | 15 | 6 | 10 | 17 | 11

2. Secondary Outcome: Number of Participants With Self-Reported Past 7-day Smoking Abstinence
Description: Number of participants that self-reported no cigarettes smoked in the past 7 days
Time Frame: 3 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Short, Short, Present | Short, Long, Present | Long, Short, Present | Long, Long, Present | Short, Short, Absent | Short, Long, Absent | Long, Short, Absent | Long, Long, Absent
Number analyzed (Participants) | 82 | 82 | 80 | 79 | 79 | 81 | 81 | 78
Participants | 6 | 11 | 10 | 14 | 8 | 14 | 12 | 7

3. Secondary Outcome: Proportion of Participants Who Reduced the Number of Cigarettes Smoked Per Day in Half
Description: Proportion of participants who reduced the number of cigarettes smoked per day in half
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Short, Short, Present | Short, Long, Present | Long, Short, Present | Long, Long, Present | Short, Short, Absent | Short, Long, Absent | Long, Short, Absent | Long, Long, Absent
Number analyzed (Participants) | 82 | 82 | 80 | 79 | 79 | 81 | 81 | 78
Participants | 21 | 24 | 31 | 23 | 21 | 27 | 29 | 22

4. Secondary Outcome: Proportion of Participants Who Reduced the Number of Cigarettes Smoked Per Day in Half
Description: Proportion of participants who reduced the number of cigarettes smoked per day in half
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Short, Short, Present | Short, Long, Present | Long, Short, Present | Long, Long, Present | Short, Short, Absent | Short, Long, Absent | Long, Short, Absent | Long, Long, Absent
Number analyzed (Participants) | 82 | 82 | 80 | 79 | 79 | 81 | 81 | 78
Participants | 21 | 23 | 23 | 26 | 19 | 21 | 26 | 23

5. Secondary Outcome: Proportion of Patients Who Make an Intentional Attempt to Quit Smoking
Description: Intentional attempt to quit smoking cigarettes that lasts for >=24 hours
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Short, Short, Present | Short, Long, Present | Long, Short, Present | Long, Long, Present | Short, Short, Absent | Short, Long, Absent | Long, Short, Absent | Long, Long, Absent
Number analyzed (Participants) | 82 | 82 | 80 | 79 | 79 | 81 | 81 | 78
Participants | 37 | 40 | 33 | 44 | 36 | 38 | 35 | 29

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 12 weeks after completion of first counseling session.
Description: Our trial is not an drug trial or intervention.
Arm/Group | Short, Short, Present | Short, Long, Present | Long, Short, Present | Long, Long, Present | Short, Short, Absent | Short, Long, Absent | Long, Short, Absent | Long, Long, Absent
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/82 | 0/80 | 0/79 | 0/79 | 0/81 | 0/81 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/82 | 0/80 | 0/79 | 0/79 | 0/81 | 0/81 | 0/78
Other Adverse Events (participants affected / at risk) | 0/82 | 0/82 | 0/80 | 0/79 | 0/79 | 0/81 | 0/81 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT03611881/Prot_SAP_000.pdf